CLINICAL TRIAL: NCT03551808
Title: Prophylactic Effect of Ketorolac Tromethamine on the Cystoid Macular Edema After Phacoemulsification in Diabetic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 96316
Record Dates: First submitted 2018-04-10; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-04

CONDITIONS: Cystoid Macular Edema After Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- installation of Ketorolac Tromethamine Eye Drop (Active Comparator)
  Interventions: Drug: using of Ketorolac Tromethamine Eye Drop
- not receiving placebo (No Intervention)

INTERVENTIONS:
Drug: using of Ketorolac Tromethamine Eye Drop — using of Ketorolac Tromethamine Eye Drop one day before the surgery in each 8 hours and continue it for 4 weeks after the surgery
  Arms: installation of Ketorolac Tromethamine Eye Drop

SUMMARY:
The aim of the study is determining the prophylactic effect of ketorolac tromethamine drop 0.5% eye drop on the functional and anatomical ocular characteristics of the diabetic patients after the phacoemulsification surgery. Cystoid macular edema (CME) is a ocular disease which the retinal thickness is increased by 30 % incidence at least or the visual acuity is decreased to 20/40 according to clinical definition. Ketorolac tromethamine is an non steroidal anti inflammatory medication which is used for treatment and Prophylactic for CME. Teh aim of this study is prophylactic effect of ketorolac tromethamine on choroidal and retinal thickness after Phacoemulsification in Diabetic Patients. In this randomized clinical trial, 102 eyes of 102 diabetic patients were included. All patients were undergone phacoemulsification surgery at Torfeh Eye Hospital between September 2015 and January 2017. To evaluate the prophylactic effect of ketorolac tromethamine topical eye drop, all cases were asked to apply it one day before the s:surgery in each 8 hours and continue it for 4 weeks after the surgery. Controls were not received placebo. All study population were examined using Snellen visual acuity chart, enhanced depth imaging optical coherence tomography (EDI-OCT). All patients were followed at 6, 12 and 24 weeks after the cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients (type II) with cataract
* Eligible patients at age range of 20 to 95 years old

Exclusion Criteria:

* Cases with a diabetic macular edema
* proliferative diabetic retinopathy
* history of intravitreal injection of bevacizumab and macular photocoagulation prior three months to the cataract surgery
* glaucoma
* refractive errors of more than ±6 diopters
* history of previous ocular surgery
* ocular pathological disorders
* history of systemic diseases
* history of medications which have a side effect on the retinal thickness
* patients with a follow up of less than 6 months
* individuals with any intraoperative complications will be excluded from this study.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Best Corrected visual acuity | 24 weeks after the surgery
  Snellen visual acuity chart

SECONDARY OUTCOMES:
retinal and choroidal thickness | 24 weeks after the surgery
  enhanced depth imaging optical coherence tomography (EDI-OCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran, Iran

REFERENCES:
- [Derived] Mohammad-Rabei H, Sabbaghi H, Emamverdi M, Karimi S, Ramezani A, Nikkhah H, Kheiri B, Yaseri M, Sheibani K, Bahreini R. The effect of topical ketorolac tromethamine on macular thickening after phacoemulsification in diabetic patients. BMC Ophthalmol. 2023 Jul 14;23(1):320. doi: 10.1186/s12886-023-03077-y. PMID 37452330